CLINICAL TRIAL: NCT02728336
Title: MRI Assessment of Patient Suitability for Cardiac Resynchronization Therapy (CRT)
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01686
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Resynchronization Therapy; Magnetic Resonance Imaging (MRI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Failure Patients (Active Comparator): patients who are scheduled to undergo clinically ordered CRT for heart failure complicated by dyssynchrony
  Interventions: Procedure: Cardiac MRI
- Control (Active Comparator): 20 matched control subjects
  Interventions: Procedure: Cardiac MRI

INTERVENTIONS:
Procedure: Cardiac MRI

SUMMARY:
The goals of this project are to: 1) explore the potential use of magnetic resonance imaging (MRI) data for improved prediction of response to cardiac resynchronization (CRT), and 2) use the MRI-derived data together with a computer model of the cardiovascular system to study the relative roles of different factors in the mechanical effects of dyssynchrony in failure, and in the response (or lack thereof) to CRT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18 and over scheduled by conventional criteria (symptomatic impairment of cardiac function with broadened QRS) for clinical CRT procedures at NYULMC.
* Normal kidney function as determined by GFR levels.

Inclusion Criteria for Controls

* Normal kidney function as determined by GFR levels
* No significant cardiovascular disease or risk factors.

Exclusion Criteria:

* electrical implants such as cardiac pacemakers or perfusion pumps
* ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants
* ferromagnetic objects such as jewelry or metal clips in clothing (which will be removed)
* pre-existing medical conditions including a likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Derivation of score of patient suitability for CRT | 4 Years
  Binary logistic regression and receiver operating characteristic curve (ROC) analyses will be used to assess the utility of baseline (pre-CRT) MRI-derived measures, alone and in combination, for the prediction of response to CRT.

CONTACTS AND LOCATIONS:
Overall Officials: Leon Axel, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States